CLINICAL TRIAL: NCT02376166
Title: M-RePoRT: Metformin - Rising PSA Remote Trial
Brief Title: Metformin for Rising PSA Remote Trial
Acronym: M-RePoRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Matthew Galsky (Other)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Associate Professor, Medicine, Hematology and Medical Oncology, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GCO 14-0472
Record Dates: First submitted 2015-02-24; First posted 2015-03-03 (Estimated); Results first posted 2017-12-22 (Actual); Last update posted 2017-12-22 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin (Experimental): 850 mg PO once daily for 4 weeks
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — 850 mg PO twice daily for the remainder of the study period (the dose of metformin will be increased to the 850 mg PO twice daily dose in the absence of grade > 1 toxicities)
  Other Names: Glucophage

SUMMARY:
Clinical trials are critical to informing the care of patients with cancer. However, only 3-5% of patients with cancer enroll in clinical trials. Poor accrual to trials has major implications with regards to the pace of progress, the cost of clinical cancer research, and the generalizability of results. The investigators have recently shown in an analysis of 7,776 cancer clinical trials registered on clinicaltrials.gov that approximately 20% of cancer clinical trials fail to complete enrollment at all; the most often cited reason was poor accrual.

Prior research has identified barriers to cancer clinical trial accrual that can be generally categorized in the domains of availability, awareness, and acceptance. Much attention has been paid to the barriers involvement awareness and acceptance - however, trial availability is likely a "rate limiting step". This pilot study is the first in a series of planned steps to attempt to shift the current paradigm of "bringing patients to trials" to "bringing trials to patients." With the integration of telemedicine visits, the investigators aim to decrease the burden of participation for patients, begin to address geographic barriers, and ultimately improve trial accrual. In this study, men with biochemically recurrent prostate cancer (a rising PSA after definitive local therapy) will receive the antidiabetic drug, metformin. Patients will require a single on-site visit for study enrollment. The remainder of the 6 month study will be conducted via a HIPPA secure telemonitoring system (monthly visits conducted via telemedicine with tablet computers provided to each patients).

DETAILED DESCRIPTION:
Men with an isolated PSA recurrence after local therapy are an ideal population for the evaluation of novel therapies given the minimal disease burden, generally indolent natural history, and patients' preference to avoid the adverse effects of androgen deprivation therapy. Metformin has shown anti-prostate cancer activity in preclinical models and cohort studies. Metformin, a biguanide oral antihyperglycemic agent, abrogates hyperinsulinemia in individuals with and without diabetes and has shown promising anti-prostate cancer activity in preclinical models, epidemiologic studies, and retrospective cohorts. Several epidemiologic/retrospective studies have shown that metformin has a positive impact on overall survival among men with prostate cancer.

These nonclinical and clinical studies have led to calls for prospective studies of metformin in patients with prostate cancer. This is a pilot telemedicine study of metformin in patients with a rising PSA ("biochemical recurrence") after definitive local therapy for prostate cancer.

The current study is supported by the following rationale:

* A large proportion of clinical trials close prematurely due to poor accrual.
* Geographic inaccessibility is a barrier to clinical trial participation.
* Metformin is a safe and inexpensive medication that has demonstrated anti-prostate cancer activity in nonclinical and epidemiologic studies. Importantly, metformin has been shown to be safe in non-diabetic patients (e.g., patients with polycystic ovary disease) and does not cause hypoglycemia.
* Use of novel technologies may facilitate clinical trial accrual and minimize the burden of participation for patients. Ultimately, these approaches may also decrease the cost of drug development and increase the pace of progress.

In the absence of prohibitive toxicities or disease progression (defined in 4.4), patients may continue treatment for the 6-month study period. This study will include a baseline visit for study enrollment at Mount Sinai. The remainder of the visits will be telemedicine visits conducted using secure video conferencing.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate. (*in situations where pathology reports documenting prostate cancer are no longer available such as when the initial biopsy or prostatectomy was performed in the remote past, a documented history of prior prostate cancer and prostate cancer treatment in prior medical records will be sufficient)
* Biochemical disease progression after radical prostatectomy and/or radiation therapy (external-beam radiation therapy and/or brachytherapy), and no radiographic evidence of metastases.

  * Men with history of radical prostatectomy are required to have baseline PSA > 0.5 ng/mL (Prior treatment with neoadjuvant, adjuvant, or salvage radiation therapy is allowed, again, with screening PSA greater than or equal to 0.5 ng/mL required for eligibility).
  * Men treated with primary radiation therapy are required to have baseline PSA ≥ 1.0 ng/mL above their post radiation nadir for men who were treated with primary radiation therapy (external beam and/or brachytherapy). Men who had primary radiation therapy followed by salvage prostatectomy are eligible if screening PSA is greater than or equal to 0.5 ng/mL.
  * Men with previous neoadjuvant adjuvant hormone therapy are eligible if testosterone level at screening is non-castrate (≥ 50 ng/dl). Men previously treated with intermittent hormonal therapy are also eligible if level of testosterone at screening is non-castrate (≥ 50 ng/dl).
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).
* Subjects must have normal organ as defined below:

  * AST(SGOT)/ALT(SGPT) less than or equal to 1.8 X institutional upper limit of normal
  * Serum bilirubin ≤ ULN (except for subjects with Gilbert's Disease who are eligible despite elevated serum bilirubin level)
  * Creatinine ≤ 1.5 mg/dL and/or creatinine clearance > 60 ml/min
* English speaking

Exclusion Criteria:

* Concurrent use of other investigational agents or other prostate cancer therapies (e.g., androgen deprivation therapy)
* Currently taking metformin, sulfonylureas, thiazolidinedione, insulin, or other antidiabetic drugs for any reason.
* Known hypersensitivity or intolerance to metformin
* Condition associated with increased risk of metformin-associated lactic acidosis:

  * New York Heart Association Class III or IV Heart Failure
  * Intake of 3 or more alcoholic beverages per day
  * Known history of lactic acidosis

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Result] Galsky MD, Shahin M, Jia R, Shaffer DR, Gimpel-Tetra K, Tsao CK, Baker C, Leiter A, Holland J, Sablinski T, Mehrazin R, Sfakianos JP, Acon P, Oh WK. Telemedicine-Enabled Clinical Trial of Metformin in Patients With Prostate Cancer. JCO Clin Cancer Inform. 2017 Nov;1:1-10. doi: 10.1200/CCI.17.00044. PMID 30657386

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin
Started | 15
Completed | 12
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Discontinued metformin early | 2

BASELINE CHARACTERISTICS:
Arm/Group | Metformin
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 68 [57 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Gleason Score [Median (Full Range); unit: units on a scale] — A system of grading prostate cancer tissue based on how it looks under a microscope. Gleason scores range from 2 to 10 and indicate how likely it is that a tumor will spread. A low Gleason score means the cancer tissue is similar to normal prostate tissue and the tumor is less likely to spread; a high Gleason score means the cancer tissue is very different from normal and the tumor is more likely to spread.
  units on a scale | 7 [6 to 9]
Primary Treatment [Count of Participants; unit: Participants]
  Radical prostatectomy | 12
  Radiation therapy | 3
Years from local therapy to study enrollment [Median (Full Range); unit: years] | 5.9 [1.2 to 16.0]
Baseline PSA [Median (Full Range); unit: ng/mL] | 4.1 [0.52 to 31.7]
One-way driving distance to study center [Median (Full Range); unit: miles] | 63.2 [2.4 to 146]
One-way driving time to study center [Median (Full Range); unit: minutes] | 71 [12 to 147]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Completed All Telemedicine Visits
Description: Feasibility will be defined as completion of all telemedicine visits by > 2/3 of enrolled patients (unless treatment discontinued early for toxicity or disease progression).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Metformin: 850 mg PO once daily for 4 weeks Metformin: 850 mg PO twice daily for 5 months (the dose of metformin will be increased to the 850 mg PO twice daily dose in the absence of grade > 1 toxicities)
Arm/Group | Metformin
Number analyzed (Participants) | 15
Participants | 12

2. Secondary Outcome: Percentage of Participants With Stable PSA Levels at 6 Months as Defined by a <20% Change
Description: Percent of patients with 6-month PSA stable 20% change at 6 months as compared to baseline
Time Frame: baseline and 6 month
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 12
Participants | 7

3. Secondary Outcome: Adherence With Metformin as Measured by Electronic Pill Adherence Monitoring
Description: Adherence with metformin as measured by electronic pill adherence monitoring. Patients were provided with an electronic medication dispenser/medication adherence monitoring device. The device provided audible and visual reminders to proceed with drug dosing and was equipped with a cellular modem that registers a signal to a cloud-based database each time a patient accessed his or her study medication. However, the size and shape of the metformin pills caused the device to malfunction frequently, which led patients to access the pills from the device manually; the data, therefore, could not be used for analysis.
Time Frame: 6 months
Arm/Group | Metformin
Number analyzed (Participants) | 0

4. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 1
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "I would participate in a clinical trial in the future".
Time Frame: 6 months
Population: 2 patients did not complete the questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 10
  Agree | 3
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

5. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 2
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "I would participate in a telemedicine clinical trial in the future".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 9
  Agree | 4
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

6. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 3
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "The time commitment required for participation in this trial was not overly burdensome".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 11
  Agree | 2
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

7. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 4
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "Participation in this trial did not disrupt my work or other activities".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 11
  Agree | 2
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

8. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 5
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "I found it easy to use the telemonitoring tablet computer".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 5
  Agree | 2
  Neither agree nor disagree | 0
  Disagree | 4
  Strongly disagree | 2

9. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 6
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "This telemedicine approach eases the travel burden for participation in clinical trials for patients".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 10
  Agree | 3
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

10. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 7
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "This telemedicine approach eases the financial burden of participation in clinical trials for patients".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 11
  Agree | 2
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

11. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 8
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "My local physician was adequately informed about my participation in this trial (if applicable)".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 11
  Agree | 2
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

12. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 9
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "I felt I was monitored sufficiently closely while enrolled in this trial".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 11
  Agree | 2
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

13. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 10
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "I would recommend participation in a telemedicine clinical trial to other patients".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 11
  Agree | 2
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

14. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 11
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "I would participate in a clinical trial where the entire trial was conducted remotely without requiring any visits to the study center".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 8
  Agree | 3
  Neither agree nor disagree | 1
  Disagree | 0
  Strongly disagree | 1

15. Secondary Outcome: Patient Satisfaction as Measured by a Patient Satisfaction Survey Question 12
Description: Patient satisfaction with the remote clinical trial experience as measured by a patient satisfaction survey - "I felt that I was able to communicate well with the study team, even though most contact was through the tablet computer video instead of in person".
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin
Number analyzed (Participants) | 13
Participants
  Strongly agree | 12
  Agree | 1
  Neither agree nor disagree | 0
  Disagree | 0
  Strongly disagree | 0

16. Secondary Outcome: Urgency to Have a Bowel Movement Episodes
Description: Quality of LIfe as measured by a modified RAND 36-Item Health Survey. Ist reported outcome - Number of episodes of urgency to have a bowel movement
Time Frame: 6 months
Measure: Number; unit: episodes
Arm/Group | Metformin
Number analyzed (Participants) | 13
episodes
  No problem | 4
  Very small problem | 4
  Small problem | 1
  Moderate problem | 1
  Big problem | 0

17. Secondary Outcome: Increased Frequency of Bowel Movements
Description: Quality of LIfe as measured by a modified RAND 36-Item Health Survey. Ist reported outcome - Number of episodes of Increased frequency of bowel movements
Time Frame: 6 months
Measure: Number; unit: episodes
Arm/Group | Metformin
Number analyzed (Participants) | 13
episodes
  No problem | 6
  Very small problem | 3
  Small problem | 0
  Moderate problem | 1
  Big problem | 0

18. Secondary Outcome: Episodes of Watery Bowel Movements
Description: Quality of LIfe as measured by a modified RAND 36-Item Health Survey. 2st reported outcome - Number of episodes of watery bowel movements
Time Frame: 6 months
Measure: Number; unit: episodes
Arm/Group | Metformin
Number analyzed (Participants) | 13
episodes
  No problem | 4
  Very small problem | 3
  Small problem | 2
  Moderate problem | 1
  Big problem | 0

19. Secondary Outcome: Episodes of Flatulence
Description: Quality of LIfe as measured by a modified RAND 36-Item Health Survey. 3rd reported outcome - Number of episodes of flatulence
Time Frame: 6 months
Measure: Number; unit: episodes
Arm/Group | Metformin
Number analyzed (Participants) | 13
episodes
  No problem | 8
  Very small problem | 1
  Small problem | 1
  Moderate problem | 0
  Big problem | 0

20. Secondary Outcome: Episodes of Bloating
Description: Quality of LIfe as measured by a modified RAND 36-Item Health Survey. 4th reported outcome - Number of episodes of bloating
Time Frame: 6 months
Measure: Number; unit: episodes
Arm/Group | Metformin
Number analyzed (Participants) | 13
episodes
  No problem | 8
  Very small problem | 1
  Small problem | 1
  Moderate problem | 0
  Big problem | 0

21. Secondary Outcome: Episodes of Nausea
Description: Quality of LIfe as measured by a modified RAND 36-Item Health Survey. 5th reported outcome - Number of episodes of nausea
Time Frame: 6 months
Measure: Number; unit: episodes
Arm/Group | Metformin
Number analyzed (Participants) | 13
episodes
  No problem | 8
  Very small problem | 1
  Small problem | 0
  Moderate problem | 1
  Big problem | 0

22. Secondary Outcome: Episodes of Vomiting
Description: Quality of LIfe as measured by a modified RAND 36-Item Health Survey. 6th reported outcome - Number of episodes of vomiting
Time Frame: 6 months
Measure: Number; unit: episodes
Arm/Group | Metformin
Number analyzed (Participants) | 13
episodes
  No problem | 10
  Very small problem | 0
  Small problem | 0
  Moderate problem | 0
  Big problem | 0

ADVERSE EVENTS:
Arm/Group | Metformin
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metformin (N=15)
Dehydration (General disorders) | 1 (1) — Dehydration from anorexia and nausea requiring hospitalization. Resolved with discontinuation of metformin and intravenous hydration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin (N=15)
Abdominal cramps (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Anorexia (General disorders) | 2
Bloating (Gastrointestinal disorders) | 2
Consitipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 12
Dyspepsia (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 6
Flatulence (Gastrointestinal disorders) | 1
Indigestion (Gastrointestinal disorders) | 1
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Nausea (General disorders) | 1
Pain (General disorders) | 1
Queasiness (General disorders) | 1
Vomiting (General disorders) | 1
Weight loss (General disorders) | 1

LIMITATIONS AND CAVEATS:
One limitation was the need for a single onsite enrollment visit, which likely still represents a significant geographic barrier to trial accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes